CLINICAL TRIAL: NCT03705988
Title: A Double-blind, Randomized, Sham-controlled Study of Cranial Electrotherapy Stimulation as an Add-on Treatment for Tic Disorders in Children and Adolescents(SCATT)
Brief Title: A Study of Cranial Electrotherapy Stimulation as an Add-on Treatment for Tic Disorders (SCATT)
Acronym: SCATT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20182032-1
Record Dates: First submitted 2018-09-29; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Tic Disorder, Childhood
Keywords: Tic disorders; Tourette Syndrome; Cranial Electrotherapy Stimulation; CES
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm (Experimental): Participants will receive 40 sessions in 4 weeks, for twice daily on weekdays from Monday to Friday. Each session will be performed for 30 minutes. The current intensity will be adjusted continuously from 500 μA~2mA.
  Interventions: Device: Cranial Electrotherapy Stimulation(CES)
- Sham Arm (Sham Comparator): Participants will receive 40 sessions in 4 weeks, for twice daily on weekdays from Monday to Friday. Each session will be performed for 30 minutes. The current intensity will be adjusted lower than 100 μA.
  Interventions: Device: sham Cranial Electrotherapy Stimulation( sham CES)

INTERVENTIONS:
Device: Cranial Electrotherapy Stimulation(CES) — Cranial electrotherapy stimulation (CES) has been known as a kind of noninvasive treatment, which applies pulsed, weak electrical current to head through two electrodes that placed on the earlobes. The current intensity could be adjusted continuously from 500 μA~2mA.
  Arms: Intervention Arm
Device: sham Cranial Electrotherapy Stimulation( sham CES) — Cranial electrotherapy stimulation (CES) has been known as a kind of noninvasive treatment, which applies pulsed, weak electrical current to head through two electrodes that placed on the earlobes. The sham CES devices were identical to the active device, except the ear clip electrodes emit electricity intensity of lower than 100 μA.
  Arms: Sham Arm

SUMMARY:
Tic disorders is recognized as a neuropsychiatric disease. The treatments of tic disorders include drug therapy, psychotherapy and physical therapy. As a non-invasive therapy, cranial electrotherapy stimulation(CES) is approved to have few side effects and applied in various areas, especially in psychiatric diseases. However, up to now there have been no results about the effects of CES in the treatment of tic disorders.The investigators hope CES could offer a useful approach for treating tic disorders.

DETAILED DESCRIPTION:
The investigators will conduct a randomized, double-blind, sham-controlled trial to determine the efficacy of CES as an add-on treatment for tic disorders (SCATT). The study will be conducted at an outpatient, single-center academic setting. A total of 100 patients aged 6 to 17 years with tic disorders and lack of clinical response to 4 weeks' pharmacotherapy will be enrolled. Patients will be randomly into 2 groups and given 4 weeks' treatment, including 40 daily 30-minute sessions of active CES(500μA~2mA) or sham CES(lower than 100μA) on weekdays. Change in Yale Global Tic Severity Scale (YGTSS) is considered to be the primary outcome. The secondary outcome is the changes in Clinical Global Impression (CGI) and Hamilton Anxiety Scale (HAMA). Assessments will be performed at baseline, week 2, week 4 and week 8. Adverse events(AE) will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-17 years old
* Diagnosed with TD, according to Intentional Classification of Diseases (ICD-10) criteria, currently in a phase of exacerbation.
* Presented to be lack of response to medication after 4 weeks of treatment

Exclusion Criteria:

* Physical illnesses, such as cholera, hepatolenticular degeneration, myoclonic epilepsy, drug-induced extrapyramidal symptoms and organic diseases
* Substance dependence and abuse
* Severe psychiatric disease, such as depression, bipolar disorder, schizophrenic disease,
* Risk for suicide or attempted suicide
* Researchers think that the patient is not suitable for the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Yale Global Tic Severity Scale (YGTSS) score | 8 weeks
  Change in Yale Global Tic Severity Scale (YGTSS) at baseline and week 2, 4, 8. The YGTSS is applied by means of a semistructured interview with multiple informants (generally, the parents) who assess the child's tics over a period of at least one week.

SECONDARY OUTCOMES:
Changes in Clinical Global Impression (CGI) score | 8 weeks
  Change in Clinical Global Impression (CGI) between groups at baseline and week 2, 4, 8.
Changes in The Hamilton Rating Scale for Anxiety (HAM-A) score | 8 weeks
  Change in The Hamilton Rating Scale for Anxiety (HAM-A) at baseline and week 2, 4, 8.
  The HAM-A consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scores range from 0 to 56 where 14-17 indicates mild anxiety, 18-24 indicates moderate anxiety and scores of 25 and over indicate severe anxiety.
adverse effects | 8 weeks
  Any adverse event notified spontaneously by the subject, or observed by the research team will be recorded on the form designed for this purpose. The researcher will classify the intensity of adverse events in accordance with the following scale: Mild: some discomfort experienced but not such as to interrupt normal daily activity.
  Moderate: sufficient discomfort to reduce or notably affect normal daily activity. Severe: provoking incapacity to work or perform normal daily activity.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Huaning, Doctor, Study Chair — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Wu Wenjun, Master, Study Director — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Xi Min, Master, Principal Investigator — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Wu Di, Master, Principal Investigator — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Yan Qinghong, Bachelor, Principal Investigator — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.

IPD SHARING:
Plan to Share IPD: No
Patients are all children and adolescents. We decided not to share IPD to protect the personal information of the patients.

REFERENCES:
- [Background] Sukhodolsky DG, Woods DW, Piacentini J, Wilhelm S, Peterson AL, Katsovich L, Dziura J, Walkup JT, Scahill L. Moderators and predictors of response to behavior therapy for tics in Tourette syndrome. Neurology. 2017 Mar 14;88(11):1029-1036. doi: 10.1212/WNL.0000000000003710. Epub 2017 Feb 15. PMID 28202705
- [Background] Eapen V, Cavanna AE, Robertson MM. Comorbidities, Social Impact, and Quality of Life in Tourette Syndrome. Front Psychiatry. 2016 Jun 6;7:97. doi: 10.3389/fpsyt.2016.00097. eCollection 2016. PMID 27375503
- [Result] Schmitt R, Capo T, Boyd E. Cranial electrotherapy stimulation as a treatment for anxiety in chemically dependent persons. Alcohol Clin Exp Res. 1986 Mar-Apr;10(2):158-60. doi: 10.1111/j.1530-0277.1986.tb05064.x. PMID 3521373
- [Result] Ferdjallah M, Bostick FX Jr, Barr RE. Potential and current density distributions of cranial electrotherapy stimulation (CES) in a four-concentric-spheres model. IEEE Trans Biomed Eng. 1996 Sep;43(9):939-43. doi: 10.1109/10.532128. PMID 9214809
- [Result] Childs A. Cranial electrotherapy stimulation reduces aggression in a violent retarded population: a preliminary report. J Neuropsychiatry Clin Neurosci. 2005 Fall;17(4):548-51. doi: 10.1176/jnp.17.4.548. PMID 16387997
- [Result] Bystritsky A, Kerwin L, Feusner J. A pilot study of cranial electrotherapy stimulation for generalized anxiety disorder. J Clin Psychiatry. 2008 Mar;69(3):412-7. doi: 10.4088/jcp.v69n0311. PMID 18348596
- [Result] Feusner JD, Madsen S, Moody TD, Bohon C, Hembacher E, Bookheimer SY, Bystritsky A. Effects of cranial electrotherapy stimulation on resting state brain activity. Brain Behav. 2012 May;2(3):211-20. doi: 10.1002/brb3.45. PMID 22741094
- [Result] Kirsch DL, Nichols F. Cranial electrotherapy stimulation for treatment of anxiety, depression, and insomnia. Psychiatr Clin North Am. 2013 Mar;36(1):169-76. doi: 10.1016/j.psc.2013.01.006. PMID 23538086
- [Result] Barclay TH, Barclay RD. A clinical trial of cranial electrotherapy stimulation for anxiety and comorbid depression. J Affect Disord. 2014 Aug;164:171-7. doi: 10.1016/j.jad.2014.04.029. Epub 2014 Apr 21. PMID 24856571
- [Result] Qiao J, Weng S, Wang P, Long J, Wang Z. Normalization of Intrinsic Neural Circuits Governing Tourette's Syndrome Using Cranial Electrotherapy Stimulation. IEEE Trans Biomed Eng. 2015 May;62(5):1272-80. doi: 10.1109/TBME.2014.2385151. Epub 2014 Dec 22. PMID 25546850